CLINICAL TRIAL: NCT05785247
Title: Evaluating the Implementation of Head and Neck Cancer E-health Study (ENHANCE): A Hybrid Type 2 Implementation-effectiveness Study to Evaluate a Cancer Support App in Patients With Head and Neck Cancer
Brief Title: ENHANCE - Evaluating the Implementation of Head and Neck Cancer E-health
Acronym: ENHANCE
Status: Active, not recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 321026
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Head and Neck Neoplasms
Keywords: implementation; digital health; ehealth; self-management; cancer support apps
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The NHS Long Term Plan has an ambition to provide patients with digital services and tools to give them more control over their own health and care. Guy's Cancer Centre in London (UK) is offering patients with head and neck cancer (HNC) the use of a smartphone cancer support app. Few studies have evaluated the best way to implement apps to support patients with cancer, nor explored how they could help patients to self-manage. This is a hybrid implementation-effectiveness study to evaluate the implementation of a cancer-specific self-management app currently being used at Guy's Cancer Centre. The purpose of the study is to assess the following: (1) key implementation outcomes, including acceptability and usability; (2) barriers and facilitators to patients and staff using the app; (3) the effectiveness of the app to support patients to self-manage during treatment for HNC.

Eligible participants include patients being treated for HNC, and their oncology clinical team. The study will be conducted at Guy's Cancer Centre, a comprehensive cancer centre in London, UK.

The study will employ mixed methods. Data collection will involve questionnaires to measure the acceptability and usability of the app, and routinely collected patient-reported outcome measures. In addition, a sub-sample of participants will take part in semi-structured interviews to explore how the app was used and views about the implementation process. Findings from this study will identify barriers and facilitators to using the app and context about how it may help patients to self-manage their condition. These findings will help to refine ongoing development of digital cancer services. Findings will inform the development of recommendations for the integration of digital health in cancer services that can be shared with Cancer Alliances across the UK.

ELIGIBILITY:
Inclusion Criteria:

* Individuals currently undergoing treatment for head and neck cancer, under the care of an oncologist, or
* Health professionals involved in the care of patients using the app, or involved in the implementation of the app

Exclusion Criteria:

* Individuals who are not able to speak or understand English, due to no translation services available
* Patients with ECOG Performance Status Scale level 3 or 4 at baseline

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals currently undergoing treatment for head and neck cancer or (b) the healthcare staff involved in their care, who are currently using the app as part of local service improvement initiative
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Adoption | End of study, 12 months
  % of patients and staff to adopt the app

SECONDARY OUTCOMES:
Health-related quality of life | after 8 weeks of app use
  Measured with EORTC QLQ C30 score
Health-related quality of life | after 8 weeks of app use
  Measured with EORTC QLQ HN43 score
Health Service Resource Utilization | After 8 weeks of app use or at EOT
  Including unplanned hospital attendance (and length of inpatient stay), A&E visits, urgent care use, unscheduled clinic visits, self-reported by patients at end of each treatment cycle or week and calculated as group proportions over the entire course of treatment.
Patient and staff experience | after 8 weeks of app use
  Qualitative interviews and focus groups will explore experience of app use in different groups (patients and staff)
Symptom Severity | Baseline (within 1 week before treatment starts). Mid-way throughout treatment (week 3-6 - dependent on treatment type) and EOT (around week 6-12)
  Symptom severity will be measured using Common Terminology Criteria for Adverse Events (CTCAE). CTCAE is a multidimensional clinician-reported assessment that evaluates physical and psychological symptoms according to their frequency, severity and distress/bother to the person in the past week.
Clinician acceptability | End of study or 6 months since implementation of the app
  Using the Normalization Measurement Development questionnaire to assess clinicians' acceptance and perceptions of normalising behaviour into routine practice
User/Satisfaction, System Usability | 8 weeks of app use
  post-implementation mHealth app usability questionnaire (patients and staff) designed to assess users' perceived satisfaction with mobile health applications. Questionnaire items are organized into scales, with each scale assumed to measure an attribute related to usability.
Acceptability, appropriateness, and feasibility | after 8 weeks of app use
  Qualitative interviews with app users to explore experience of app usage as part of routine care

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lei, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
anonymised quantitative data will be deposited in the King's Open Research Data System (KORDS), at King's College London